CLINICAL TRIAL: NCT06793020
Title: Use of an Integrated Mathematical Model for the Diagnosis, Treatment and Outcome Assessment of Septic Cardiomyopathy
Brief Title: Diagnosis, Treatment, and Outcome Assessment of Septic Cardiomyopathy Using an Integrated Mathematical Model
Status: Recruiting | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Tomas Jovaisa, Prof, Vilnius University
Other Study IDs: 2024-3-1574-1032; 2024/3-1574-1032 (Other: Vilnius Regional Biomedical Research Ethics Comittee)
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-08

CONDITIONS: Septic Cardiomyopathy
Keywords: Septic cardiomyopathy; Sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate whether a new integrated mathematical model can improve the accuracy of diagnosing septic cardiomyopathy and predicting clinical outcomes in adult patients with suspected septic cardiomyopathy. The study aims to determine whether the integrated mathematical model enhances diagnostic accuracy and improves the prediction of clinical outcomes in these patients.

DETAILED DESCRIPTION:
This multicenter, prospective observational study will enrol adult patients treated for sepsis or septic shock in the intensive care unit (ICU). Eligible patients will be identified based on predefined inclusion and exclusion criteria and enrolled in the study after obtaining informed consent. The primary transthoracic echocardiography will be performed within 48 hours of enrollment to gather detailed echocardiographic data, while key hemodynamic measurements will be recorded simultaneously.

A second transthoracic echocardiography will be conducted within 10 days of the initial evaluation. This follow-up assessment will occur during continued ICU care after discontinuation of vasopressor therapy or during hospitalization in the general ward, depending on the patient's clinical progression. The echocardiographic and hemodynamic parameters from both the initial and follow-up evaluations will be input into a mathematical formula designed to integrate these data into a single cardiovascular estimate. This integrated model will then be used to assess its ability to predict patient outcomes.

Following hospital discharge, patients will be followed for up to one year. During this period, a long-term follow-up assessment will be conducted, during which patients will complete the SF-36 quality of life questionnaire. This follow-up will assess patients' overall health, functional status, frequency of healthcare visits, and need for nursing care. These data will provide insights into the long-term impact of sepsis and septic cardiomyopathy on survivors beyond the acute phase of their illness.

This study will evaluate whether the use of an integrated model that combines clinical parameters with echocardiographic measurements can improve the accuracy of diagnosing septic cardiomyopathy and provide valuable predictions of clinical outcomes. Additionally, the study will assess the course of septic cardiomyopathy and its impact on one-year follow-up outcomes, including patient quality of life. A broadly applicable diagnostic approach could allow for timely treatment adjustments, reduce the burden of sepsis-related complications, and improve overall patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Sepsis according to SEPSIS-3 criteria:
* Suspected/confirmed infection and
* SOFA (Sequential Organ Failure Assessment) score ≥ 2 or qSOFA score ≥ 2;
* Septic shock according to SEPSIS-3 criteria:
* Sepsis is diagnosed and
* Vasopressor infusion is used to maintain a mean arterial pressure (MAP) ≥ 65 mmHg and
* Lactate > 2 mmol/l;
* Cardiovascular support requirement for norepinephrine > 0.1 mcg/kg/min infusion;
* Signed informed consent form (ICF);

Exclusion Criteria:

* Individuals under 18 years of age;
* Has uncompensated cardiovascular disease:
* Cardiogenic shock;
* Congenital heart disease;
* Heart failure NYHA functional class IV;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for sepsis or septic shock in the Intensive Care Units of two university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of septic cardiomyopathy when comparing a new clinical-echocardiographic model with the standard diagnostic method (left ventricular ejection fraction). | From enrollment to the end of one-year follow-up.
  Incidence of septic cardiomyopathy, evaluated by comparing the diagnostic accuracy of a new clinical-echocardiographic model with the standard method, left ventricular ejection fraction (LVEF) measurement. The study will determine whether the new model improves the diagnosis of septic cardiomyopathy in patients with sepsis or septic shock.

SECONDARY OUTCOMES:
Assessing the severity of septic cardiomyopathy and determining the severity grade. | From enrollment to the end of one-year follow-up.
  This will be done by applying clinical and echocardiographic data to the integrated mathematical model, which will then categorize the severity of the condition into predefined severity grades. The assessment aims to provide a more nuanced understanding of the diseases impact on cardiac function and to validate the models ability to stratify patients based on the severity of their condition.
Length of intensive care unit and hospital stay | Intensive care unit days spent per patient: within 60 days following intensive care unit admission. Hospital days spent per patient: from admission up to 30 days.
  Total cumulative number of days spent in intensive care unit and hospital
Mortality | Within 1 year of inclusion
  Mortality during intensive care unit stay, in hospital and at 1 year
Recovery of cardiac function | Within 30 days of inclusion
  Changes in the integrated mathematical model during hospitalization
Long-term health and functional outcomes | Within 1 year of inclusion
  Heath-related quality of life assessed by Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). Assessment of changes in functional capacity, number of visits to healthcare facilities, and the need for nursing care.

CONTACTS AND LOCATIONS:
Locations (2):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- University Clinical Centre of the Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No